CLINICAL TRIAL: NCT05975697
Title: The EFFECT of FUNCTIONAL ELECTRICAL STIMULATING on PHYSICAL ACTIVITY and QUALITY of LIFE in PATIENTS with PARALIS AFTER THROMBECTOMY: a RANDOMIZED CONTROLLED STUDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ceylan Kisial, PhD student, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CK-01
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-08

CONDITIONS: Thrombectomy
Keywords: Thrombectomy; FES; PHYSICAL ACTIVITY; LIFE QUALITY; Nursing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Divided into two groups as experimental and control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is planned to be double-blind, and the patient and the evaluating physician will not know which patient is in the study group and which patient is in the control group. The walkers and the physiotherapist will not be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group to be applied FES (Experimental): FES treatment to the deltoid, triceps, extensor carpi radialis muscles for a total of 10 sessions, 30 minutes twice a day (in the morning and in the evening), for 5 days after the first 24th hour after the thrombectomy procedure in the experimental group patients (Program duration is 15 minutes and resting time is 15 minutes). minutes) will be applied.
  Interventions: Other: Experimental group to be applied FES
- control group (No Intervention): In the control group patients; From the first 24 hours after the thrombectomy procedure, the routine of the clinic (such as not performing a non-pharmacological procedure) is applied for 5 days, and no other procedure will be performed.

INTERVENTIONS:
Other: Experimental group to be applied FES — In the first 24 hours after the thrombectomy procedure, the relatives of the patients in the experimental and control groups who meet the inclusion criteria will be informed by the researcher and their consent will be obtained.
  FES treatment to the deltoid, triceps, extensor carpi radialis muscles for a total of 10 sessions, 30 minutes twice a day (in the morning and in the evening), for 5 days after the first 24th hour after the thrombectomy procedure in the experimental group patients (Program duration is 15 minutes and resting time is 15 minutes). minutes) will be applied.Patient information form (Appendix 1), Fugl-meyer upper extremity motor assessment scale (Appendix-2) and Quick DASH (Arm, Shoulder and Hand Injury Questionnaire Short Form) (Appendix-3) were given to both groups within the first 24 hours after the thrombectomy procedure. ) will be applied. All patients will be re-evaluated before and on the 5th day after treatment.
  Arms: Experimental group to be applied FES

SUMMARY:
It is planned as a randomized controlled intervention study to determine the effect of functional electrical stimulation (FES) on physical activity and quality of life in patients with paralysis after thrombectomy.

DETAILED DESCRIPTION:
Thrombectomy is an interventional radiology procedure, and especially a method used endovascularly, and is the removal of a blood clot formed in arteries and veins (Yıldırım, 2023). Timely restoration of cerebral blood flow using reperfusion therapy is the most effective maneuver to save uninfarcted ischemic brain tissue (Jadhav at al., 2018). As the benefit of reperfusion decreases over time, one of the most common complications as a result of increasing ischemic areas is paralysis (Powers at al., 2019).

Paralysis often leads to significant impairment in upper extremity function and is associated with reduced quality of life in all domains except mobility (Franceschini at al., 2010). More than half of the patients may become partially or completely dependent on others in daily activities (Aşiret at al., 2013; Coban., 2013; Rahmani Anaraki at al., 2013; Kheirollahi at al., 2013). However, few patients achieve full functional recovery, and this deficiency impairs the performance of all physical activities, including self-care and social activities (Kwakkel at al., 2003). Different therapeutic methods are used to prevent or reduce the long-term deterioration of the upper extremities in patients undergoing thrombectomy (Vafadar at al., 2015). Among these therapeutic methods, non-pharmacological methods are much easier to learn, safe and without definite contraindications (Howlett at al., 2015).

According to the studies reviewed, functional electrical stimulation (FES) is a non-pharmacological method, which is a device that electrically stimulates motor neurons to improve motor functions aimed at stimulating the nerves of weakened muscles (Lynch at al., 2008; Niu, at al., 2022). Transcutaneous electrodes offer an easy and fast treatment option because they are non-invasive (Eraifej at al., 2017).

As a result of the literature review, FES (Bolton at al., 2004; Howlett at al., 2015; Meilink at al., 2008; Vafadar at al., 2015; Van Peppen at al., 2004) has proven its effectiveness in the rehabilitation of the lower extremity after thrombectomy. , and there is no clarity about the effectiveness of FES in upper extremity rehabilitation (Stroke rehabilitation in adults. Published June 2013. Accessed 1 Jan 2016). This is partly due to methodological limitations (Howlett at al., 2015; Vafadar at al., 2015) or the outdated nature of some existing studies (Bolton at al., 2004; Meilink at al., 2008; Van Peppen at al., 2004). ). It was also highlighted by a recent Cochrane review that required a current review and meta-analysis of randomized controlled trials (RCTs) on electrical stimulation (Pollock at al., 2014). The most recent recent systematic review found a significant improvement in motor outcomes with the upper extremity FES (Howlett at al., 2015).

In this context, FES application in our country is one of the functional applications of nurses to correct the activity with the doctor and to exercise management (https://www.resmigazete.gov.tr/eskiler/2011/04/20110419-5.htm). In our study, we aimed to base the effect of functional electrical stimulation (FES) on physical activity and quality of life in patients with paralysis after thrombectomy, and to form a source for current and similar studies.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Thrombectomy procedure was performed,
* Glasgow Coma Score (GCS) > 12 after thrombectomy
* Able to communicate,
* Having upper extremity paralysis,
* No pacemaker, advanced spasticity and muscle atrophy, peripheral lesions, osteoporosis, skin irritation and obesity,
* No skin and peripheral circulation problems,
* Patients whose relatives gave consent to the research.

Exclusion Criteria:

* Patients who did not comply with the sampling criteria and who developed complications that caused brain damage during the study (convulsions, mental disorder/delirium, vomiting, tremor, myoclonus) and whose relatives did not approve of the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Rating Scale (FMRS) | 5 days
  To assess motor function, the Fugl Meyer Rating Scale (FMRS) considers the upper extremity in 3 parts. These parts are shoulder-elbow-forearm, (upper arm) wrist and hand. The score evaluation is 36 points for the upper arm, 10 points for the wrist and 14 points for the hand evaluation. In the evaluation of coordination and speed, the maximum total score of the upper extremity is 66, out of 6 points.

SECONDARY OUTCOMES:
Quick DASH (Arm Shoulder and Hand Injury Questionnaire Short Form) | 5 days
  The questionnaire consists of 11 questions, and the difficulties of the patients during their daily living activities are examined. Each answer is scored from 1 to 5 on a Likert scale, from best to worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No